CLINICAL TRIAL: NCT06552325
Title: Integrating Brief Narrative Therapy in Low Barrier Clinics to Enhance HIV Prevention
Brief Title: Walk-in Therapy in Low Barrier Primary Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Lydia Chwastiak, Professor, Psychiatry and Behavioral Sciences, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00018557; 3P30MH123248-03 (NIH)
Record Dates: First submitted 2024-08-10; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Mental Health Issue; Hiv; Substance Use
Keywords: Houselessness; Brief narrative therapy; Implementation outcome; Integrated care; Reach
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Session Narrative Therapy Intervention (Experimental): A single narrative therapy session with a trained licensed behavioral health provider will be offered to patients at [Blinded] low-barrier clinics.
  Interventions: Behavioral: Single Session Narrative Therapy

INTERVENTIONS:
Behavioral: Single Session Narrative Therapy — The proposed single session narrative therapy intervention has been widely implemented in walk-in therapy clinics in Ontario Province, Canada. In these clinics, 60-minute psychotherapy sessions, informed by narrative therapy, are available on a walk-in basis. The therapist collaborates with a patient to co-develop a useful and meaningful focus for the session and then engages the patient in conversation that is respectful but shifts their way of thinking about the presenting problem. The therapist highlights and documents the patient's values and skills and works with the patient to create an action plan. If the therapist identifies additional treatment needs, the patient is offered an external referral to specialty mental health services.
  Other Names: Brief Narrative Therapy

SUMMARY:
The goals of the current research are to adapt an effective walk-in psychotherapy clinic intervention for the context of low-barrier primary care; and conduct a pilot implementation study in two low-barrier primary care clinics that are based in a community organization that is a drop-in center for people experiencing homelessness in North Seattle.

DETAILED DESCRIPTION:
Interactions between the multiple health threats of mental illness, substance use, and social vulnerabilities (homelessness, poverty) represent a syndemic that perpetuates the HIV epidemic. Mental health and substance use disorders have been shown to increase HIV risk behaviors and to have a negative impact on adherence to PrEP. Unhoused individuals face both individual-level (stigma, limited social support, and psychiatric symptoms) and structural-level (poverty, unstable housing, limited transportation, cost of medical care) barriers to healthcare. Walk-in clinics are designed to address these barriers to traditional primary care and provide immediate access to services when they are needed. King County WA has funded four low-barrier primary care clinics since 2018 as a key component of the King County EHE Plan. Data from these clinics suggest that untreated mental disorders are a critical barrier to engagement in low-barrier primary care. Integrated care models in which trained mental health specialists deliver evidence-based mental health care in primary care settings increase access to care by providing mental health treatment where people are already seeking care. Integrated care improves mental health outcomes, and models are feasible to implement even in very low resource settings. Walk-in counseling clinics throughout the province of Ontario, Canada, have implemented a single session narrative therapy intervention to increase access to mental health care. In this model, therapists use a single-session approach to help clients identify issues, recognize and build on their strengths and develop an action plan. Narrative approaches create a non-pathologizing, collaborative, and competency-oriented way of addressing mental health needs. Given the unpredictability of follow-up in walk-in primary care, a single session narrative approach can make the most of every single session, providing pragmatic therapeutic conversations to people when they need it and support coping, reduce feelings of isolation, and increase sense of validation. The goals of the current study are 1) to develop a single-session narrative therapy intervention to increase access to mental health care among people experiencing homelessness; and 2) conduct a 4-month pilot implementation trial of the adapted intervention in two low-barrier primary care clinics in North Seattle.

ELIGIBILITY:
Patient Inclusion Criteria:

* Will have completed at least one therapy appointment at the [Blinded] clinics
* Ability to provide informed consent
* Ability to complete the interview or questionnaire in English

Patient Exclusion Criteria:

* Inability to provide informed consent
* Need for urgent mental health treatment (e.g., imminent risk of harm to self or others, acute withdrawal requiring medical detoxification)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Reach | Up to 4 months
  Number and representativeness of patients (with respect to gender, race/ethnicity, current substance use) who have ≥1 session with the therapist (compared to full clinic populations).

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Chwastiak, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: Yes
Research subject's de-identified data will be shared through the National Institute of Mental Health Data Archive (NDA).
Time Frame: Data will made available in alignment with the first data submission date required by the National Institute of Mental Health Data Archive.
Access Criteria: Summary information on the data shared in NDA is available in the NDA Query Tool without the need for an NDA user account. To request access to record-level human subject data, a Data Access Request must be submitted.